CLINICAL TRIAL: NCT01902563
Title: Osteopathic Approach Into Neonatology Ward: the NE-O Model
Status: Available | Type: Expanded Access
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NE-O-prot
Record Dates: First submitted 2013-07-10; First posted 2013-07-18 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: The Focus of the Study is to Provide a Guideline on Osteopathic Approach in Treating Hospitalized Newborns.
Keywords: osteopathic manipulative treatment; newborns; preterm infants; procedures
MeSH Terms: interventions — Manipulation, Osteopathic

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment

SUMMARY:
Background Several studies have shown the effect of osteopathic manipulative treatment on neonatal care in reducing length of stay, gastrointestinal problems, clubfoot complications and improving cranial asymmetry of infants affected by plagiocephaly. Despite several results obtained, there is still lack of standardized osteopathic evaluation and treatment procedures for newborns recovered in neonatal intensive care unit (NICU).

The aim of this research is to provide a guideline on osteopathic approach in treating hospitalized newborns. Specific evaluation tests and treatments have been developed to tailor osteopathic method according to preterm and term infants' needs, NICU environment, medical and paramedical assistance.

ELIGIBILITY:
Inclusion Criteria:

* newborn admitted to neonatal intensive care unit
* informed consent signed from parent or legal guardian

Exclusion Criteria:

* post surgery patients

Ages: 29 Weeks to 40 Weeks | Sex: All
Age Groups: Child